CLINICAL TRIAL: NCT06014281
Title: An Internet-administered Randomized Control Trial to Examine the Effects of Regular, Brief Meditation Practice on Mental Health and Well Being
Brief Title: Examining the Effects of Regular Brief Internet-based Meditation Practice on Mental Health and Well Being
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Institute for Meditation and Inner Harmony (Unknown); Feldman Foundation CA (Unknown)
Responsible Party: Principal Investigator, Manish Saggar, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68784
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meditation group (Experimental): Baseline to week 8:
  Subjects will be trained to meditate for 10 minutes daily, and several measures (questionnaires, cognitive tests, and physiological measurements) will be obtained to assess the efficacy of daily meditation practice on mental health and well being. Focused-attention meditation technique will be used to train participants. Specifically the SOS meditation technique will be employed.
  Week 8 to week 16:
  Subjects will self report if they choose to continue SOS meditation and several measures (questionnaires, cognitive tests, and physiological measurements) will be obtained to assess the impact of continued meditation practice on mental health and well being.
  Interventions: Behavioral: SOS Meditation
- Waitlist control (Experimental): Baseline to week 8:
  Subjects will be place in a control group which receives no intervention. However, several measures (questionnaires, cognitive tests, and physiological measurements) will be obtained to assess baseline mental health and well being scores.
  Week 8 to week 16:
  Subjects will be trained to meditate for 10 minutes daily, and several measures (questionnaires, cognitive tests, and physiological measurements) will be obtained to assess the efficacy of daily meditation practice on mental health and well being. Focused-attention meditation technique will be used to train participants. Specifically the SOS meditation technique will be employed.
  Interventions: Behavioral: SOS Meditation

INTERVENTIONS:
Behavioral: SOS Meditation — Focused-attention meditation technique will be used to train participants, specifically the SOS meditation technique. The SOS meditation technique is an easy-to-learn approach where participants are instructed to dissociate their attention from physical awareness, thoughts, and emotions by mentally slowly repeating a calming word or phrase (chosen by the participant themselves).
  SOS Meditation Instructions:
  * Close your eyes very gently, in a relaxed way, as you do when we go to sleep
  * Your attention should be fully alert. Try not to put any strain on your eyes or try to look up.
  * Focus your eyes about eight to ten inches into the field of darkness in front of you on the horizontal plane
  * Mentally repeat the (chosen) calming word
  * Sit lovingly and calmly to see what comes up, as if you were watching a movie screen and waiting to see what appears on it.

SUMMARY:
The study will examine the effects of online meditation training on stress and anxiety in healthy participants. It will also examine the dose-response relationship between the amount of daily focused attention meditation practice and established mental health outcome measures.

DETAILED DESCRIPTION:
This is a 16-week study with an 8-week meditation intervention, with a requirement of a minimum of 10 minutes of meditation practice each day. This study will recruit ~200 healthy subjects (18+ years) with no current or previous diagnosis of psychiatric or neurological disorders who are interested in learning about meditation but don't have long-term experience with meditation. Half of the participant pool will be randomly assigned to the meditation intervention, and the other half will get the wait-list control assignment. The control group will later receive its intervention, likely a few weeks after the completion of the active group's intervention. A focused-attention meditation technique (SOS meditation) will be used to train participants.

Changes in participants' physiological markers (e.g., HRV, physical activity, respiration rate, sleep quality) will be evaluated using passive activity monitoring devices (e.g., Fitbit). Intervention-related changes in mental health will be assessed using web-based mental health and well-being surveys. Improvements in cognitive functioning will be assessed using web-based psychological tasks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to follow basic instructions for prescreening and scheduling
* Compliant with investigator instructions during the consent process and participation in the study
* Is not already a regular meditation practitioner

Exclusion Criteria:

* Age <18
* People with a current diagnosis of psychiatric or neurological disorders
* Be in current psychiatric treatment or medications
* Hospitalized for psychiatric disorders in the past year or so.
* Regular and long-term meditation practitioners
* Non-English speaking
* Non-USA mailing address to receive the activity tracker device
* Vision or hearing impairment severe enough to interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Generalize Anxiety Disorder Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Anxiety as measured using Generalize Anxiety Disorder Questionnaire
Change in Pittsburgh Sleep Quality Index Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Sleep Quality measured using Pittsburgh sleep quality index (PSQI)
Change in Mind Wandering Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Mind wandering measured using the Mind Wandering Questionnaire
Resting Heart Rate | Daily (from baseline to week 8 for arm 1 and from week 8 to week 16 for arm 2)
  Daily obtained from Activity Tracker wrist band
Heart Rate Variability | Daily (from baseline to week 8 for arm 1 and from week 8 to week 16 for arm 2)
  Daily obtained from Activity Tracker wrist band
Change in Stroop Test Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Using the Stroop test, which measures the average reaction time between incongruent and congruent trials
Change in N-back Test Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Using the N-back test is a memory task where participants must remember letters from N trials ago.

SECONDARY OUTCOMES:
Change in Stress Scale Measure Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Stress measured using Perceived Stress Scale measure
Change in Depression Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Depression measured using Patient Health Questionnaire
Change in Quality of Life Scale Measures Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Quality of life measured using Quality of Life Scale measures
Change Social Connectedness Scale-Revised Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Social Connectedness measured using Social Connectedness Scale-Revised
Change in Rumination Reflection Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Rumination and reflection scales measured using Rumination Reflection Questionnaire
Change in Brief Strengths Scale Questionnaire Score | Twice (Baseline and week 8 for arm 1 and week 8 and week 16 for arm 2)
  Strengths scale measured using Brief Strengths Scale measures individuals' Temperance Strength, Intellectual Strength, and Interpersonal Strength.
Change in Sleep Quality Measure | Daily (from baseline to week 8 for arm 1 and from week 8 to week 16 for arm 2)
  Daily obtained from Activity Tracker wrist band

CONTACTS AND LOCATIONS:
Overall Officials: Manish Saggar, PhD, Principal Investigator — Stanford University
Locations (1):
- Dept. of Psychiatry, Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No